CLINICAL TRIAL: NCT06722053
Title: Effects of Integrative Sensory-Supported Virtual Reality and Gamified Digital Breastfeeding Education on Mothers' Breastfeeding Success, Self-Efficacy and Adaptation
Brief Title: Integrated Sensory Supported Virtual Reality and Gamified Digital Breastfeeding Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ipek turhan (Other)
Responsible Party: Sponsor-Investigator, ipek turhan, PhD student, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ErciyesU-SBF-IT-02
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Feeding
Keywords: breasfeeding; virtual reality; gamification
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: There are two intervention groups and one control group.
Who Masked: Outcomes Assessor
Masking Description: The person administering the surveys will not know which group the participants are in, so blinding will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group 1 (Other): Receiving breastfeeding skills training and gamified digital foundation training with virtual reality.
  Interventions: Other: virtual reality and digital education
- intervention group 2 (Other): With virtual reality breastfeeding skills training, gamified digital-based breastfeeding training will be provided, and in addition, there will be a lemon oil scent in the environment during virtual reality breastfeeding skills training and in the postpartum period.
  Interventions: Other: virtual reality and digital education; Other: virtual reality and digital education and lemon scent
- control group (No Intervention): No training or intervention will be applied and will receive the hospital's standard treatment, care and education.

INTERVENTIONS:
Other: virtual reality and digital education — Breastfeeding education through virtual reality and digital education
  Arms: intervention group 1; intervention group 2
Other: virtual reality and digital education and lemon scent — virtual reality and digital education and lemon scent inhalation
  Arms: intervention group 2

SUMMARY:
Breastfeeding is the most ideal form of nutrition that concerns the health of mother and baby. The World Health Organization (WHO) recommends that breastfeeding should be started within the first hour after birth. Although breastfeeding has many benefits, research shows that breastfeeding rates are not at the desired level. Breastfeeding self-efficacy, success and adaptation become important to increase breastfeeding rates. In order to provide these components related to breastfeeding, breastfeeding education must be given starting from prenatal period. Education methods have taken different forms in line with the developing technology and the needs of the generation. WHO states that information and communication technology is an opportunity to support breastfeeding. Virtual reality and online learning applications also positively affect learning. New teaching methods, which are increasingly used today, make learning easier and can be used easily in virtual environments. Providing learning by doing in a realistic environment is important for successful breastfeeding and gaining breastfeeding skills and competence. In order to gain breastfeeding skills, the mother can experience breastfeeding during pregnancy using virtual reality technology. While breastfeeding skills are gained through virtual reality, information about breastfeeding can be provided through gamified digital training. With the game, the student actively participates in education. Active participation of the student in gamification ensures that knowledge becomes permanent. It is thought that the effect of the integrative sense can be used to facilitate postpartum remembering of these trainings.

DETAILED DESCRIPTION:
Breastfeeding is the key to sustainable development. The second and third goals of the Sustainable Development Goals, a strategy plan to increase the development levels of countries by 2030 at the United Nations (UN) Sustainable Development Summit, are directly related to breastfeeding. The second of the Sustainable Development Goals is "Eradicate Hunger", while the third article directly related to breastfeeding is "Healthy Individuals". Breastfeeding is the only practice that will prevent hunger and malnutrition in the newborn and infancy period. Increasing breastfeeding can make positive contributions to the health of newborns, infants and children . Breastfeeding is the most ideal form of nutrition regarding the health of mothers and infants. The World Health Organization (WHO) recommends that breastfeeding should be initiated within the first hour after birth . Although breastfeeding has many benefits, studies show that breastfeeding rates are not at the desired level. The UNICEF 2019 report states that breastfeeding within the first hour following birth is 43%, and exclusive breastfeeding for the first six months is 41% . The Turkey Demographic and Health Survey 2018 breastfeeding and breastfeeding data show that 98% of children born in the last two years in Turkey were breastfed for any period of time. The percentage of breastfeeding within the first hour after birth is 71. Breastfeeding results are not at the targeted level due to the mother's attitude, lack of knowledge, incorrect breastfeeding methods, breast problems such as breast fullness, breast abscess, nipple pain and mastitis. Educating and supporting women about breastfeeding is very important in terms of increasing breastfeeding rates . For this reason, breastfeeding education should be started before birth and postpartum problems should be detected and resolved early. Receiving breastfeeding education positively affects breastfeeding success. WHO states that information communication technology is an opportunity to support breastfeeding. With the developing technology in recent years, mobile applications and the internet have become a source of health information. The development of mobile health technology increases patients' health knowledge and awareness and reduces the workload in the health field . It is seen that traditional methods cannot be successful in education due to reasons such as the increasing population, the distance of health institutions, and the inability of health workers and patients to spare time for health education. However, web-based training has advantages such as using visual and auditory methods together, updating the training content, not requiring transportation to the hospital, reaching different people simultaneously, reducing workload and costs . With developing technology, breastfeeding training has begun to be provided with technology-based methods. Since the learner is usually in a passive role in traditional training, critical thinking, problem-solving skills and the sense of living in the moment may not develop . Although the level of knowledge and learning is higher in breastfeeding training where visual materials are used compared to plain narration, breastfeeding skills cannot be developed and competence cannot be achieved . However, new teaching methods, which are increasingly used today, make learning easier and can be easily used in virtual environments. At the same time, virtual reality and online learning applications also positively affect learning . Recently, gamification has been used in online learning trainings to make trainings more interesting. Gamification is the process of presenting information by turning it into a game. Gamified teaching makes the learning process more attractive and increases motivation. With the game, the student actively participates in the training. The active participation of the student in gamification ensures that the knowledge becomes permanent. Studies have shown that web-based trainings increase breastfeeding self-efficacy and that continuing with breastfeeding support is also useful and up-to-date. Web-based trainings are interesting and effective compared to formal education. Combining these trainings with gamification will increase motivation and permanence of knowledge. However, breastfeeding is a psychomotor skill . Evidence-based guidelines recommend practical trainings to support breastfeeding . Learning by doing in a realistic environment

ELIGIBILITY:
Inclusion Criteria:

* literate,
* healthy (no systemic/chronic disease, diagnosed psychiatric or neurological disease, no risky pregnancies, etc.)
* primiparous pregnant women with singleton pregnancies,
* planning to breastfeed,
* having an internet-connected smart phone/tablet/computer and being able to use it actively,
* competent enough to play games and having no problems with their hands, no breast problems that would make breastfeeding difficult (indentation, missing nipple, sore nipple, etc.),
* no vision, hearing or communication problems,
* pregnant women who are not allergic to lemon or lemon oil

Exclusion Criteria:

* the occurrence of a situation that prevents sucking
* the baby is not healthy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since breastfeeding is done by women, the study will be conducted with women.
Enrollment: 105 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale | first day postpartum and thirtieth day postpartum
  The Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, in 2003, Dennis reduced the scale to 14 items and developed the Breastfeeding Self-Efficacy Scale Short Form. The Turkish validity and reliability of the Breastfeeding Self-Efficacy Scale Short Form was conducted by Aluş Tokat and Okumuş (2010). This scale evaluates how competent mothers feel about breastfeeding. The 14-item scale includes a 5-point Likert-type assessment consisting of the options Not at all sure (1), Not very sure (2), Sometimes sure (3), Sure (4) and Very sure (5). The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score obtained from the scale indicates a high perception of breastfeeding self-efficacy. This scale can be applied in both the antenatal and postnatal periods. The difference between the antenatal form and the postnatal form of the scale is the use of the expression "future tense" in the scale items.
LATCH Diagnostic Scale | first day postpartum
  The LATCH Breastfeeding Assessment Tool was created in 1986 by resembling the APGAR scoring system in terms of scoring method. The scale was developed to objectively diagnose breastfeeding, identify breastfeeding problems, plan training, create a common language among healthcare professionals, and be used in research. The scale, which is quick and easy to evaluate, consists of five evaluation criteria. Each item is evaluated between 0 and 2 points. The total possible score is 10 and there is no cut-off point. As the score increases, it is understood that breastfeeding success is high. .
Breastfeeding Adaptation Scale | first day postpartum and thirtieth day postpartum
  The Breastfeeding Adaptation Scale was developed by Sun Hee Kim (2009). The Turkish validity and reliability were made by Dinçel and Özdilek (2021). Scale items were rated with a 5-point Likert (1 point: Strongly disagree, 2 points: Disagree, 3 points: Undecided, 4 points: Agree, 5 points: Strongly agree). The items in the 6th sub-dimension of the scale, "breastfeeding discomfort", are reverse coded. The score that can be obtained from the scale varies between 27-135. An increase in the total score indicates a high level of breastfeeding adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: ipek turhan, master, Principal Investigator — Kayseri City Hospital
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study has not started, it is not planned to be shared at the moment for the confidentiality of the study idea.